CLINICAL TRIAL: NCT02597894
Title: Feasibility of Repeat Targeted Biopsies in Patients Undergoing High-Dose-Rate Prostate Brachytherapy
Brief Title: Targeted Biopsies in Determining Response in Patients With Prostate Cancer Undergoing High-Dose-Rate Brachytherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: P. I. left the Institution. Study never opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-000360; NCI-2015-01737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID562 (Other: Jonsson Comprehensive Cancer Center); 15-000360 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-11-02; First posted 2015-11-05 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2017-04

CONDITIONS: Stage III Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostate biopsy (Other): Patients undergo two biopsies, the first at baseline before start of ADT and the second two months later during brachytherapy.
  Interventions: Procedure: Biopsy of Prostate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies targeted biopsies in determining response in patients with prostate cancer undergoing high-dose-rate brachytherapy (a type of radiation therapy in which radioactive material sealed in needles, seeds, wires, or catheters is placed directly into or near a tumor). Studying tumor tissue obtained before and after treatment may help doctors understand changes in a pathway that looks at how deoxyribonucleic acid (DNA) is repaired after it is damaged and to see if there are differences in the prostate tissue prior to and after starting androgen deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate feasibility of obtaining adequate tumor tissue from an intra-prostatic index lesion prior to the start of androgen deprivation therapy (ADT) and again at the time of high-dose-rate (HDR) brachytherapy.

SECONDARY OBJECTIVES:

I. Use immunohistochemistry to stain cells pre-ADT and post 2 months of ADT for markers of non-homologous end joining and DNA double strand breaks using the following markers: Ku70, Ku80, DNA-dependent protein kinase catalytic subunits (PKCs), gamma-histone family, member X (H2AX).

OUTLINE:

Patients undergo biopsy at baseline before start of ADT and during brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma of the prostate
* National Comprehensive Cancer Network (NCCN) high risk disease (cT3 or Gleason score 8-10 or prostate specific antigen [PSA] > 20)
* Not currently on ADT
* Magnetic resonance imaging (MRI) or transrectal doppler ultrasound demonstrating at least one target lesion
* Karnofsky performance status (KPS) >= 70 or Eastern Cooperative Oncology Group (ECOG) = 2
* Understands the trial and procedure and is willing and able to sign the informed consent form

Exclusion Criteria:

* Patient is unable to receive high dose rate prostate brachytherapy
* Patient is unable to have a MRI or transrectal ultrasound
* Refusal to sign the informed consent
* Patients who are participating in a concurrent treatment protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in DNA damage repair pathways | Two months
  The prostate biopsy sample at baseline and at the time of brachytherapy (approximately two months later) will be examined to determine if prostate cancer is in the core and if at least 20% of the core has prostate cancer in it.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Kamrava, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States